CLINICAL TRIAL: NCT00580736
Title: Optical Clearing of the Skin in Conjunction With Laser Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D., Professor Departments of Dermatology and Surgery, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20033442
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain; Nevus of Ota; Tattoos; Scars; Acne; Hypertrichosis; Sebaceous Gland Diseases
Keywords: sebaceous hyperplasia
MeSH Terms: conditions — Port-Wine Stain; Nevus of Ota; Cicatrix; Acne Vulgaris; Hypertrichosis; Sebaceous Gland Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Clearing (Experimental): Optical Clearing
  Interventions: Device: Optical Clearing

INTERVENTIONS:
Device: Optical Clearing — Optical Clearing

SUMMARY:
The research hypothesis is that topical application of a mixture of pre-polymers of polypropylene glycol and polyethylene glycol (an optical clearing agent) will reduce skin light scattering, increasing the amount of light reaching the target for diagnostic as well as therapeutic purposes.

DETAILED DESCRIPTION:
The researchers expect that application of the optical clearing agent for treatment of benign vascular lesions, tattoos, nevus of Ota, hypertrichosis, scars, acne and sebaceous hyperplasia will result in

1. decreased reflectance of the predominant color from the surface of skin (decreased red light scattering in case of benign vascular lesions, etc) as compared to the control group.
2. greater Optical Coherence Tomography a non-invasive light based imaging method imaging depth as compared to the control group.
3. greater improvement in the treatment outcome (decrease in the erythema index following laser treatment of vascular lesions as compared to the laser alone group; improved lightening of the tattoo or nevus of Ota as compared to the laser treatment alone group; significant decrease in hair re-growth as compared to laser treatment alone in patients seeking hair removal; greater improvement of scars, acne and sebaceous hyperplasia).

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* Lesion diagnoses in an area measuring 3 cm2 or more on any body site
* Apparent good health

Exclusion Criteria:

* Pregnant women
* History of cutaneous photosensitivity
* History of photodermatoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Outcome measure is to evaluate the optical clearing effects of the combination mixture of pre-polymers of polypropylene glycol and polyethylene glycol. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, M.D, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute Medical and Surgical Clinic, Irvine, California, United States